CLINICAL TRIAL: NCT04942314
Title: Practice of Treat-to-target on Pediatric Systemic Lupus Erythematosus: a Two-center Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jia Deng (Other)
Collaborators: Children's Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor-Investigator, Jia Deng, Master of medical degree, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: CHChongqingMU-2021.03.30
Record Dates: First submitted 2021-06-06; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: pediatric; SLE; treat to target
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Complete remission off therapy: 1. no clinical activity and serological activity
  2. stop taking corticosteroid and immunosuppressive drugs
  3. antimalarials allowed
- Complete remission on therapy: 1. no clinical activity and serological activity
  2. corticosteroid≤5 mg/day and immunosuppressive drugs allowed
  3. antimalarials allowed
- Clinical remission off therapy: 1. no clinical activity but serological activity allowed
  2. stop taking corticosteroid and immunosuppressive drugs
  3. antimalarials allowed
- Clinical remission on therapy: 1. no clinical activity but serological activity allowed
  2. corticosteroid≤5 mg/day and immunosuppressive drugs allowed
  3. antimalarials allowed
- Low disease activity state: (1) SLEDAI-2K ≤4, with no activity in major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, fever), and no haemolytic anaemia or gastrointestinal active involvement; (2) no new lupus disease activity compared with the previous assessment; (3) a PGA ≤1; (4) a current predni- sone (or equivalent) dose ≤7.5mg/day; and (5) well-tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.
- Not in LDAS or Remission: At the end of follow-up, the disease state of SLE children was not in LDAS or any remissions defined above.
- Never in LDAS: During the follow-up, the disease state was never get LDAS.

SUMMARY:
Treat to target (T2T) strategies have proved to be useful in several chronic disorders, including Rheumatoid Arthritis. In systemic lupus erythematosus (SLE), T2T strategy has been proposed in order to control disease activity, improve health-related quality of life, and reduce morbidity and mortality. Remission would be the main target, but a low disease activity state (LDAS) could be an acceptable alternative. However, due to SLE protean manifestations, the operational definitions of both remission and LDAS are still in progress. This clinical trial would like to assess the clinical value of T2T strategy in the treatment of children with SLE, optimize the treatment of children with SLE, andimprove the prognosis.

DETAILED DESCRIPTION:
This two-center study retrospectively analyzed the follow-up data of children with systemic lupus erythematosus (SLE) in our center (the Children's Hospital of Chongqing Medical University) and the Children's Hospital of Nanjing Medical University, grouping the patients into two observation groups-low disease activity status Group (LDAS group) and never reached low disease activity group (Never LDAS group). We would analyze the risk factors of SLE that patients cannot reach LDAS by comparing baseline data and treatment conditions of the two groups. Meanwhile, we would evaluate the SLE clinical indicators, SLE disease activity, organ damage, and disease remission state at the end of the follow-up of the LDAS group, in order to assess the clinical value of T2T strategy in the treatment of children with SLE, optimize the treatment of children with SLE, andimprove the prognosis.

ELIGIBILITY:
Inclusion Criteria:

(1）Children with SLE diagnosed by the SLICC classification criteria for systemic lupus erythematosus (2012); (2) Since diagnosed of SLE to follow-up termination, inpatient and/or outpatient follow-up at the research centers shall be carried out at least twice a year, the interval of follow-up is ≤3-6 months, and the total follow-up time is ≥1 year; (3) All children or guardians signed an informed consent file before inclusion.

Exclusion Criteria:

1. the treatment plan is unknown;
2. Excluding deaths caused by other diseases
3. follow-up was interrupted;
4. Follow-up time is less than 1 year, or interval is more than 6 months.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with SLE were diagnosed in the Children's Hospital of Chongqing Medical University and the Children's Hospital of Nanjing Medical University from January 2012 to December 2019 that meet the SLICC classification criteria for systemic lupus erythematosus (2012)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Risk factors for LDAS in children's SLE | 2021.07-2023.06
  grouping the patients into two observation groups-low disease activity status Group (LDAS group) and never reached low disease activity group (Never LDAS group). By comparing baseline data and treatment conditions of the two groups, The research would analyze the risk factors of SLE that patients cannot reach LDAS including demographic features, clinical manifestation, serologically activity, therapy at baseline.

SECONDARY OUTCOMES:
assess the clinical value of T2T strategy in the treatment of children with SLE | 2021.07-2023.06
  At the end of follow up, the LDAS group would be grouped into 6 groups including complete remission off therapy, complete remission on therapy, clinical remission off therapy, clinical remission on therapy, LDAS and not in LDAS or remisson.we would evaluate the SLE clinical indicators, SLE disease activity, organ damage, and disease remission state at the end of the follow-up of the LDAS group, in order to assess the clinical value of T2T strategy in the treatment of children with SLE, optimize the treatment of children with SLE, andimprove the prognosis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ugarte-Gil MF, Burgos PI, Alarcon GS. Treat to target in systemic lupus erythematosus: a commentary. Clin Rheumatol. 2016 Aug;35(8):1903-1907. doi: 10.1007/s10067-016-3346-2. Epub 2016 Jul 12. PMID 27406378